CLINICAL TRIAL: NCT04663308
Title: A Randomized Double-Blind Placebo-Controlled Study to Evaluate the Efficacy and Safety of Volixibat in the Treatment of Cholestatic Pruritus in Patients With Primary Sclerosing Cholangitis
Brief Title: A Study to Evaluate Efficacy and Safety of an Investigational Drug Named Volixibat in Patients With Itching Caused by Primary Sclerosing Cholangitis (PSC)
Acronym: VISTAS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VLX-301; 2020-003027-41 (EudraCT Number); 2023-505764-11-00 (Other: EUCT number)
Record Dates: First submitted 2020-11-17; First posted 2020-12-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Pruritus; PSC; Itch; Itching; Cholestasis
MeSH Terms: conditions — Cholangitis, Sclerosing; Pruritus; Cholestasis | interventions — volixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Arm 1: Volixibat 20mg (Experimental): Participants randomized to this arm will receive volixibat 20mg twice daily.
  Interventions: Drug: Volixibat
- Part 1 Arm 2: Volixibat 80mg (Experimental): Participants randomized to this arm will receive volixibat 80mg twice daily.
  Interventions: Drug: Volixibat
- Part 1 Arm 3: Placebo (Placebo Comparator): Participants in this arm will receive capsules matched to the study drug minus the active volixibat substance, twice daily.
  Interventions: Drug: Placebo
- Part 2 Arm 1: Volixibat Selected Dose 20mg (Experimental): Participants randomized to this arm will receive volixibat 20mg twice daily.
  Interventions: Drug: Volixibat
- Part 2 Arm 2: Placebo (Placebo Comparator): Participants in this arm will receive capsules matched to the study drug minus the active volixibat substance, twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Volixibat — Oral capsules, administered twice daily. Volixibat is an Ileal Bile Acid Transporter (IBAT) inhibitor.
  Other Names: SHP626
  Arms: Part 1 Arm 1: Volixibat 20mg; Part 1 Arm 2: Volixibat 80mg; Part 2 Arm 1: Volixibat Selected Dose 20mg
Drug: Placebo — Capsules matched to study drug minus active substance
  Arms: Part 1 Arm 3: Placebo; Part 2 Arm 2: Placebo

SUMMARY:
The purpose of this clinical research study is to learn more about the use of the study medicine, volixibat, for the treatment of pruritus (itching) associated with Primary Sclerosing Cholangitis (PSC), and to assess the possible impact on the disease progression of PSC.

ELIGIBILITY:
Inclusion Criteria:

1. Provide freely signed informed consent and assent (as applicable) and be willing to comply with all study visits and requirements through end of study, including the follow-up period.
2. Subjects aged ≥12 years for eligible regions; otherwise ≥18 years
3. Confirmed diagnosis of large duct or small duct PSC based on American Association for the Study of Liver Disease (AASLD) guidelines.
4. Pruritus associated with PSC as assessed by Adult ItchRO.
5. Ursodeoxycholic acid (UDCA) and anti-pruritic medication use will be allowed if meeting additional criteria.
6. Concomitant Inflammatory Bowel Disease (IBD) is allowed if meeting additional criteria.

Exclusion Criteria:

1. Pruritus associated with an etiology other than PSC
2. Evidence or clinical suspicion of decompensated cirrhosis, or a history of decompensation events
3. History of ileostomy or small bowel surgery/resection or other surgeries that may have disrupted the enterohepatic circulation
4. Evidence, history, or suspicion of other liver disease; PSC patients with AIH are not excluded.
5. Bile duct stent or percutaneous bile duct drain placement, or balloon dilatation procedure of a stricture within 12 weeks of Screening
6. Exceeding pre-defined biochemical values for alanine aminotransferase/aspartate aminotransferase (ALT/AST), estimated glomerular filtration rate (eGFR),serum creatinine (sCr), platelet count, international normalized ratio (INR) and total bilirubin
7. History of liver transplantation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in the daily itch scores using the Adult Itch Reported Outcome (Adult ItchRO) questionnaire | Baseline through to Week 28
  The Adult ItchRO is an 11-point NRS measurement of itch severity ranging from 0=no itch to 10=worst possible itch.

SECONDARY OUTCOMES:
Proportion of participants with itch response using the Adult ItchRO | Baseline through to Week 28
The incidence of adverse events | Baseline through to Week 28
Changes in serum bile acid levels | Baseline through to Week 28
Changes in alkaline phosphatase | Baseline through to Week 28
Changes in total bilirubin levels | Baseline through to Week 28
Change in Primary Sclerosing Cholangitis-Specific Patient-Reported Outcome | Baseline through to Week 28
Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) fatigue questionnaire | Baseline through to Week 28
  The PROMIS® Fatigue questionnaire is a 5-point response scale. Respondents endorse each item using a 5-point response scale: Never, Rarely, Sometimes, Often, and Always.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) sleep disturbance questionnaire | Baseline through to Week 28
  The PROMIS® Sleep Disturbance in an 8-item measure that assesses quality of sleep, sleep depth, and restoration associated with sleep. It is a 5-point response scale, the specific response options vary by items. The first 4 items use response options that range from Not at all to Very much. The next 3 items use response options that range from Never to Always. The final item assesses sleep quality ranging from Very poor to Very good.

CONTACTS AND LOCATIONS:
Locations (103):
- United States (34):
  - Southern California Research Center, Coronado, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami - Schiff Center for Liver Diseases, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Northwell Health, Manhasset, New York
  - New York University Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center - Presbyterian Hospital and Vanderbilt Clinic, New York, New York
  - University of Rochester Medical Center - Strong Memorial Hospital, Rochester, New York
  - Duke Health - Duke University Medical Center, Durham, North Carolina
  - Science 37, Inc (Remote-homebased Telemedicine), Morrisville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Einstein Healthcare Network - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Galen Medical Group, Hixson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Liver Institute At Methodist Dallas Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Liver Associates of Texas, Houston, Texas
  - University of Utah Health Care, Salt Lake City, Utah
  - Bon Secours Liver Institution of Hampton Roads Mary Immaculate Hospital Office, Newport News, Virginia
  - Richmond Community Hospital LLC, Richmond, Virginia
  - University of Washington - Harborview Medical Center, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington
- Argentina (3):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Glenny Corp S.A., Ciudad Autónoma Buenos Aires
  - Hospital El Cruce, San Juan Bautista
- Australia (5):
  - Royal Adelaide Hospital, Adelaide
  - Northern Health, Epping
  - Liverpool Hospital, Liverpool
  - Austin Health, Melbourne
  - University of the Sunshine Coast, Sippy Downs
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA), Ghent
  - University Hospital Ghent, Ghent
- Brazil (5):
  - Hospital das Clinicas da UFMG, Belo Horizonte
  - Hospital Das Clinicas Da Ufg, Goiânia
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Escola Bahiana de Medicina e Saude Publica, Salvador
  - Hospital do Rim e Hipertensao, São Paulo
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - McMaster University Hospital, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - University of Calgary, Calgary
  - London Health Sciences Centre University Hospital, London
  - McGill University Health Centre - Royal Victoria Hospital, Montreal
- France (4):
  - Centre Hospitalier Universitaire Grenoble Alpes (CHU Grenoble Alpes), Grenoble
  - Centre Hospitalier Universitaire De Lille, Lille
  - APHP-Hôpital Saint Antoine, Paris
  - CHU Bordeaux - Haut Lévêque, Pessac
- Germany (9):
  - Hannover Medical School, Hanover, Lower Saxony
  - Universitaetsklinikum Bonn, Bonn, Nordrhine-Westphalia
  - Charité Universtitätsmedizin - Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Universitatsklinikum Leipzig, Leipzig
  - Otto-von-Guericke-Universitat Magdeburg, Magdeburg
  - University Hospital Tubingen Medical Clinic, Tübingen
  - St. Josefs-Hospital Wiesbaden, Wiesbaden
- Israel (9):
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - Ein Karem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - A.O.U. Federico II, Napoli
  - Azienda Ospedale Universita Padova, Padua
- Netherlands (4):
  - Amsterdam UMC - VU Medisch Centrum (VUmc), Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud University Medical Centre (MC), Nijmegen
  - Erasmus University Medical Center, Rotterdam
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
- University Hospital Zurich, Zurich, Switzerland
- United Kingdom (11):
  - Royal Free Hospital, London, Hampstead
  - John Radcliffe Hospital, Oxford, Headington
  - Royal Victoria Hospital, Belfast
  - University Hospitals Birmingham NHS Foundation Trust - Wellcome Trust Birmingham Clinical Research Facility, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge
  - Lothian NHS Board, Edinburgh
  - St James' University Hospital Leeds Teaching Hospitals NHS Trust, Leeds
  - King's College Hospital NHS Foundation Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospital NHS Trust, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton